CLINICAL TRIAL: NCT02216422
Title: An Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 Co-administered With Ribavirin (RBV) in Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection and Cirrhosis (Turquoise-IV)
Brief Title: A Study to Evaluate Chronic Hepatitis C Virus (HCV) Infection in Cirrhotic Adults With Genotype 1b (GT1b) Infection
Acronym: Turquoise-IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-252
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection
Keywords: Chronic Hepatitis C; Hepatitis C; Hepatitis C Virus; Hepatitis C Genotype 1b; Interferon-Free
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — ombitasvir; paritaprevir; Ritonavir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombitasvir/Paritaprevir/Ritonavir plus Dasabuvir with RBV (Experimental): Ombitasvir/Paritaprevir/Ritonavir (25/150/100 mg once daily) and Dasabuvir (250 mg twice daily) co-administered with weight-based Ribavirin (RBV; twice daily) for 12 weeks
  Interventions: Drug: Ombitasvir/Paritaprevir/Ritonavir; Drug: Dasabuvir; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Ombitasvir/Paritaprevir/Ritonavir — Tablet; paritaprevir co-formulated with ritonavir and ombitasvir
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; Ritonavir also known as norvir
Drug: Dasabuvir — Tablet
  Other Names: ABT-333
Drug: Ribavirin (RBV) — Tablet

SUMMARY:
This was a multicenter study evaluating the efficacy and safety of ombitasvir/paritaprevir/ritonavir and dasabuvir co-administered with ribavirin (RBV) for 12 weeks in treatment naïve and pegylated-interferon alfa-2a or alfa-2b (pegIFN)/RBV treatment-experienced, cirrhotic HCV genotype 1b-infected adults.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety and efficacy (the percentage of participants achieving a 12-week sustained virologic response (SVR12), [HCV ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks following treatment]) of co-formulated ombitasvir, paritaprevir, and ritonavir (ombitasvir/paritaprevir/r) and dasabuvir co-administered with RBV for 12 weeks in HCV genotype 1b-infected adult participants with compensated cirrhosis. The secondary objectives of this study were to assess the number and percentage of participants with virologic failure during treatment and the percentage of participants with relapse post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, genotype 1b-infection (HCV RNA level greater than 1,000 IU/mL at Screening)
* Evidence of liver cirrhosis as confirmed by liver biopsy or Fibroscan with Child-Pugh score less than or equal to 6 at Screening
* Participant had never received antiviral treatment (including pegIFN/RBV) for hepatitis C infection (treatment-naïve participant) or had documentation of meeting one of the defined categories of a treatment-experienced participants
* Absence of hepatocellular carcinoma (HCC) as indicated by a negative ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) performed within 3 months prior to screening or a negative ultrasound at screening.
* Females must be post-menopausal, of non-child bearing potential or practicing specific forms of birth control
* Males must have been surgically sterile, or agreed to practice 2 effective methods of birth control throughout the course of the study.

Exclusion Criteria:

* Positive screen for hepatitis B Surface antigen or anti-Human Immunodeficiency virus antibody
* Evidence of current or past Child-Pugh B or C classification
* Confirmed presence of hepatocellular carcinoma
* Abnormal laboratory tests
* Participant who self-reported on average drinking more than 2 drinks per day for current drinkers
* Previous treatment with a direct acting antiviral agent (DAA) containing regimen
* History of solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando M Viani, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 participants were enrolled and all the participants completed the study. All 36 participants were analyzed for both efficacy (included all participants who received at least 1 dose of study drug (ITT)) and safety.
Period: Overall Study
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses included all participants.
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Interleukin 28B (IL28B) [Number; unit: participants]
  CC | 4
  CT | 25
  TT | 7
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: Sustained Virologic Response 12 (SVR12) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ; < 25 IU/mL) 12 weeks after the last dose of study drug. Participants with missing data were imputed as failures.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV
Number analyzed (Participants) | 36
percentage of participants | 100 [90.4 to 100.0]
Statistical Analysis 1: Comparison: Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV; Test type: Superiority or Other; Percentage of Participants = 100, 95% CI 2-sided [90.4 to 100.0] — 95% confidence interval (CI) was calculated using Wilson score method

2. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure
Description: On-Treatment Virologic Failure is defined as confirmed HCV RNA >= LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir (local minimum value) in HCV RNA [2 consecutive HCV RNA measurements > 1 log10 IU/mL above nadir] at any time point during treatment, or failure to suppress during treatment [all on-treatment values of HCV RNA >= LLOQ] with at least 6 weeks [defined as active study drug duration ≥ 36 days] of treatment.
Time Frame: Day 1 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV
Number analyzed (Participants) | 36
percentage of participants | 0 [0.0 to 9.6]

3. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post- Treatment Relapse is defined as confirmed HCV RNA >= LLOQ between end of treatment and 12 weeks after last actual dose of active study drug [up to and including the SVR12 assessment time point] for a participant with HCV RNA < LLOQ at Final Treatment Visit who completes treatment.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir With RBV
Number analyzed (Participants) | 36
percentage of participants | 0 [0.0 to 9.6]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of study drug administration to 30 days after last dose of study drug (12 weeks); SAEs were also collected from the time that informed consent was obtained until the end of the study (up to 36 weeks).
Groups:
- Ombitasvir/Paritaprevir/Ritonavir Plus: Ombitasvir/Paritaprevir/Ritonavir (25/150/100 mg once daily) and Dasabuvir (250 mg twice daily) co-administered with weight-based Ribavirin (RBV; twice daily) for 12 weeks.
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 21/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir Plus (N=36)
ANAEMIA (Blood and lymphatic system disorders) | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
ASTHENIA (General disorders) | 8
FATIGUE (General disorders) | 2
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
HEADACHE (Nervous system disorders) | 4
INSOMNIA (Psychiatric disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 5
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.